CLINICAL TRIAL: NCT05524831
Title: Kinesio Taping Versus Oromotor Training on Drooling in Children With Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar Mohamed Awaad, Scientific researcher, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003677
Record Dates: First submitted 2022-08-14; First posted 2022-09-01 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Drooling; Kinesiotape; Cerebral Palsy
MeSH Terms: conditions — Sialorrhea; Cerebral Palsy | interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: 2
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- groupA(Kinesiotape) (Experimental): kinesio tape on orbicularis oris muscle for 45 minute /3times per week for 2 successive months
  Interventions: Other: KINESIOTAPE
- group B(oromotor training) (Experimental): oromotor training for 45 minute/ 3 times per week for 2 successive months
  Interventions: Other: oromotor training

INTERVENTIONS:
Other: KINESIOTAPE — kinesiotape will be applied on orbicularis oris muscle
  Arms: groupA(Kinesiotape)
Other: oromotor training — selected oromotor training: Perioral sensory stimulation ,Tapping,Tongue pressure,Jaw exercises andIntraoral stimulation
  Arms: group B(oromotor training)

SUMMARY:
Statement of the problem :

Which is more effective for treatment of drooling in children with spastic cerebral palsy; kinesio taping or oromotor training?

Null Hypothesis:

There will be no difference between the effectiveness of kinesio taping and oromotor training on drooling in children with spastic cp.

DETAILED DESCRIPTION:
Subjects:

The Study targets the children with spastic cerebral palsy from both sexes , sample size estimation will be carried out to determine the recruited number of children ,Children participating in this study will be selected randomly from Cairo pediatric physical therapy centers to participate in this study.

Study Design:

A comparative experimental design (Prospective pre-test post-test design with 2 months follow-up evaluation) .

Children will be assessed by measuring the drooling before and after two months of receiving intervention.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of spastic cerebral palsy with drooling problem.
2. The age of the selected children will range from 4to 8 years old.
3. Severe degree of drooling according to Drooling Severity and Frequency Scale.
4. Child with good head control

Exclusion Criteria:

1. Congenital problems of mouth and soft palate such as cleft lip and palate, jaw anomalies and salivary gland pathologies.
2. Epilepsy.
3. Child receiving drugs that could affect saliva production or other treatments to control drooling just before or during the study.
4. Allergic reactions to the kinesio tape.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-12-12 (Actual); Primary Completion 2022-02-26 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
assessment of drooling severity | 2 months for each participant
  by using The 5-minute drooling quotient.it is expressed as a percentage of observed drooling episodes.
assessment of drooling severity and frequency | 2months for each participant
  by using The Drooling Severity and Frequency Scale. at severity: score 1:no drool ,score5:profuse drooling. at frequency: score 1:never drool ,score4: constant drool

CONTACTS AND LOCATIONS:
Overall Officials: Hagar Awaad, Principal Investigator — Cairo University
Locations (1):
- Faculty of physical therapy ,cairo university, Cairo, Egypt